CLINICAL TRIAL: NCT07048080
Title: (P)Rehabilitation in Older People With Osteoarthritis Undergoing Total Hip Replacement : From Physicological Mechanism to Clinical Benefits
Brief Title: Prehabilitation in Older People Undergoing Total Hip Replacement
Acronym: PREHIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Principal Investigator, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FONDECYT 1251133
Record Dates: First submitted 2025-06-17; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hip Replacement in Osteoarthritis Patients; Osteoarthritis, Hip
Keywords: hip osteoarthritis; total hip replacement; resistance exercise training; older people
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The physiotherapist performing the assessments will be blind to the intervention. The blinding will extend to the data analysis team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (P)rehabilitation Group (Experimental): Participants assigned to the (p)rehabilitation group will perform a supervised Progressive Resistance Exercise Training 2 week program for the whole body three times per week before total hip replacement surgery and for 12 weeks after. In a sub-study, the first 10 participants of (P)rehabilitation group will be included to study the effects of 2 weeks prehabilitation on tissue protein synthesis rates. A two-week deuterium oxide (2H2O or 'heavy water') loading protocol will be conducted during the two week before THR surgery to assess diurnal rates of musculoskeletal protein synthesis.
  Interventions: Behavioral: (P)rehabilitation Progresive Resistance Exercise Training; Biological: Prehabilitation Group Deuterated Water
- Usual Care Group (Other): Participants assigned to the control group will receive the usual therapy, medical monitoring, and educational lectures after surgery. No intervention is planned before total hip replacement surgery. In a sub-study, the first 10 participants of Usual Care group will be included to study the effects of 2 weeks prehabilitation on tissue protein synthesis rates. A two-week deuterium oxide (2H2O or 'heavy water') loading protocol will be conducted during the two week before THR surgery to assess diurnal rates of musculoskeletal protein synthesis.
  Interventions: Biological: Usual Care Group Deuterated Water; Other: Usual Care

INTERVENTIONS:
Behavioral: (P)rehabilitation Progresive Resistance Exercise Training — The (p)rehabilitation intervention program will be based on supervised whole-body RET performed 3 times/week before (2-week) and up to 12 weeks after surgery, with one day in-between sessions. Training will consist of a 10-min warm-up, followed by one warm-up and 4 sets on leg press, leg-extension and leg abductor machines. Upper body exercises (chest press, lat pulldown and horizontal row will be performed with 2 sets of each exercise. During the 2-week training before surgery, the workload will be increased from 70% (week 1) to 80% (week 2) of 1RM (10 repetitions in each set). After surgery, the workload will be increasing from 50% of 1RM to 80% from the last 6 weeks. All the participants included in the per-protocol analysis must complete at least 80% of the training sessions. We will take into consideration the mobility precautions so as not to dislocate the prosthesis (avoid hip flexion of 90 degrees and more; do not perform adduction exercises and hip rotations).
  Arms: (P)rehabilitation Group
Biological: Prehabilitation Group Deuterated Water — In a sub-study, the first 10 participants of the (P)rehabilitation group will be included to study the effects of 2 weeks prehabilitation on tissue protein synthesis rates. A two-week deuterium oxide (2H2O or 'heavy water') loading protocol will be conducted during the two week before THR surgery to assess diurnal rates of musculoskeletal protein synthesis. This 2H2O method enables the assessment of muscle, cartilage and bone tissue protein synthesis rates when tissue samples are collected after the 2 weeks of prehabilitation.
  Arms: (P)rehabilitation Group
Biological: Usual Care Group Deuterated Water — In a sub-study, the first 10 participants of the Usual Care group will be included to study the effects of 2 weeks prehabilitation on tissue protein synthesis rates. A two-week deuterium oxide (2H2O or 'heavy water') loading protocol will be conducted during the two week before THR surgery to assess diurnal rates of musculoskeletal protein synthesis. This 2H2O method enables the assessment of muscle, cartilage and bone tissue protein synthesis rates when tissue samples are collected after the 2 weeks of usual care.
  Arms: Usual Care Group
Other: Usual Care — Participants assigned to the usual care group will receive the usual therapy, medical monitoring, and educational lectures after surgery. No intervention is planned before total hip replacement surgery. The patient is hospitalized for surgery. At hospital discharge, the usual care group will start with standard rehabilitation (sessions: 1st month, 2-3x/week, 2nd month 1-2x/week and 3rd month 1x/month) based on mobility and strength exercises without using progressive RET with machines until 3 months after surgery.
  Arms: Usual Care Group

SUMMARY:
The goal of this clinical trial is to determine the effect of Resistance Exercise Training (RET)-based (p)rehabilitation versus usual care on skeletal muscle mass and function, as well as on underlying biological processes, in older adults undergoing elective Total Hip Replacement (THR) due to severe Osteoarthritis (OA). The main questions it aims to answer are:

* What is the effects of RET-based (p)rehabilitation versus usual care to improve muscle mass and function in patients undergoing elective unilateral THR surgery for end-stage OA?
* What is the potential of certain circulating biomarkers to predict the efficacy of the musculoskeletal system response to RET in patients with severe OA? Researchers will compare RET-based (p)rehabilitation versus usual care to see if RET works to increase skeletal muscle mass and function.

Participants in the usual care group will undergo standard rehabilitation (12 weeks post-surgery), and participants in the (p)rehabilitation group will undergo RET-based full-body (p)rehabilitation (3x/week) for 2 weeks pre-surgery and 12 weeks post-surgery.

DETAILED DESCRIPTION:
Introduction: Due to age, patients suffering from osteoarthritis (OA) experience a loss of skeletal muscle mass, strength, and functional capacity both before and after total hip arthroplasty (THA). Progressive resistance exercise training (RET) is a safe and feasible intervention before and after THA. However, the physiological and clinical effects have not been investigated on a larger scale.

Objectives: To determine the effect of RET-based (p)rehabilitation versus usual care on skeletal muscle mass and function, as well as on underlying biological processes, in older adults undergoing elective THA due to severe OA.

Materials and Methods: Seventy older adults scheduled for elective unilateral THA due to severe primary OA (usual care group: n=35, ≥60 years; (p)rehabilitation group: n=35, ≥60 years) will be included in this single-blind randomized controlled trial. Participants in the usual care group will undergo standard rehabilitation (12 weeks post-surgery), and participants in the (p)rehabilitation group will undergo RET-based full-body (p)rehabilitation (3x/week) for 2 weeks pre-surgery and 12 weeks post-surgery. MRI scans of the thigh will be taken at baseline, 24 hours before, and 12 weeks after surgery to assess the cross-sectional area of the quadriceps. On the same days, blood and muscle samples will be collected, and dual-energy X-ray absorptiometry (DEXA) will be performed. Maximum strength, muscle function/morphology, physical capacity, quality of life, performance in activities of daily living, physical activity level, hip function, nutritional status, and cognitive status will also be assessed. The occurrence of serious adverse events, hospital readmissions, infections, and complications will be considered.

In a sub-study, 20 participants (n=10 from the usual care group and n=10 from the (p)rehabilitation group) will be included to investigate the effects of 2 weeks of (p)rehabilitation on tissue protein synthesis rates. A 2-week deuterium oxide (²H₂O or "heavy water") loading protocol will be implemented in both groups during the two weeks prior to THA to assess musculoskeletal tissue protein synthesis rates. This method allows for the evaluation of the protein synthesis rate in muscle, cartilage, and bone tissue when samples are collected two weeks after the (p)rehabilitation or usual care interventions. These tissues will be collected during surgery, so no additional procedures are required from participants. In addition to determining the effects of RET on protein synthesis rates in tissues relevant to musculoskeletal health, the association between protein synthesis rates and long-term clinical outcomes will also be explored.

Expected Results: It is hypothesized that 14 weeks (2 weeks pre- and 12 weeks post-surgery) of progressive RET-based (p)rehabilitation will increase muscle mass and function to a greater extent than usual care, which is based on mobility and strength exercises without progressive machine-based RET. Additionally, RET will induce an increase in protein synthesis rates in muscle, cartilage, and bone tissues through the activation/inhibition of established signaling pathway markers (Akt, mTOR, S6(K), 4E-BP1, MAFbx, MuRF1). Furthermore, it is hypothesized that the increase in protein synthesis rate in these tissues will be associated with specific circulating biomarkers of musculoskeletal health (including CTX-II, COMP, CTX-I, OC, PIIINP, S1) and will indicate gains in muscle mass and functional improvements in the progressive RET group compared to the usual care group.

These findings will define the efficacy of progressive RET-based rehabilitation in increasing muscle mass and clinical outcomes in older adults with severe hip OA undergoing THA. Better maintenance or even increases in muscle mass and strength enhance independence, prolong health, aid recovery from illness, and reduce the burden on healthcare services. This information will have a beneficial impact on the fields of exercise physiology, orthopedics, and aging for future interventions at local, regional, national, and international levels.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged from 60 y and over.
* 18.5 < BMI < 40 kg/m2.
* Individuals on waiting list to undergo a unilateral elective surgery for Total Hip Replacement due to primary severe Osteoarthritis.

Exclusion Criteria:

* Individuals with severe OA in the contralateral hip.
* Individuals who has been performing regular RET (2 or more times per week) in the previous 6 months.
* Individuals who smoke.
* Significant psychiatric or neurological disorders, with the use of acetylcholinesterase inhibitors, and untreated mood disorders or depressive pathology.
* Neuromuscular or mobility disorders that prevent safe resistance training (debilitating arthritis, spasticity/rigidity, and paralysis), along with untreated metabolic disorders (such as uncontrolled systemic hypertension).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Taken into consideration the sex distribution of patients undergoing THR surgery (i.e., more women than men), we aim to include a minimum of 18 women per group.
Enrollment: 70 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in Cross-Sectional Area of Quadriceps measured via MRI - Scanning after resistance exercise training | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention in both groups
  Anatomic CSA of the quadriceps muscle will be assessed in the study by MRI scanning at baseline, after 2 weeks of prehabilitation and after 12 weeks of rehabilitation for all participants. On the obtained MRI images, muscle tissue will be defined by threshold values of 0-100 Hounsfield Units, and the quadriceps muscle will be selected by manual tracing using ImageJ software (version 1.45d, National Institute of Health, Maryland, USA). All analyses will be performed by one investigator blinded to participant coding.
Change in Protein Synthesis Rates (MPS) on Muscle, Bone and Cartilage measured via tissue samples after resistance exercise training. | The assessment will be conducted 2 weeks before surgery and during the surgery.
  All tissue samples (muscle, cartilage and bone) will be collected through surgical excision in the sub-study, except for the vastus lateralis muscle which will be collected from the middle region of the vastus lateralis during the surgical procedure. Conventional muscle biopsy samples of the vastus lateralis will be collected to assess MPS rates and compare this between the intervention and usual care group, as well as to provide a reference to the synthesis rates of the various musculoskeletal tissues obtained during surgery. Hereafter, samples will be freed from any visible blood, immediately frozen in liquid nitrogen, and will be stored at -80°C until subsequent analysis (38). Intramuscular free and bound 2H-Alanine enrichment will be analyzed by gas-chromatography mass spectrometer (GC-MS; Agilent 5975C MSD & 7890A GC, Wilmington, DE).

SECONDARY OUTCOMES:
Change in functional capacity measured via Short Physical Performance Battery (SPPB) after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  The functional capacity is assessed through the Short Physical Performance Battery (SPPB).
Immunodetection of protein synthesis markers in tissue sample 2 weeks before surgery, during surgery and after resistance exercise training. | The assessments will be conducted with the samples obtained 2 weeks before surgery, during surgery and after 12-week intervention.
  Muscle biopsies will be obtained from the middle region of the vastus lateralis muscle. In short, skin and muscle fascia will be locally anesthetized using 1% xylocaine (except during surgery as patient is already anesthesized). After 10 minutes a small incision will be made in skin and fascia after which the biopsy needle will be introduced in the muscle to obtain small muscle samples (total ± 150 mg). Biopsy samples from all tissues will be used to perform Western Blot and PCR analyses. Specifically, (phosphorylated) protein and mRNA expression of several proteins/genes from protein synthesis (Akt, mTOR, S6(K), 4E-BP1) and degradation (MAFbx, MuRF1) pathways will be assessed according to standard procedures. In addition, potential fiber type-specific alterations in muscle fiber size, myonuclear and/or satellite cell content will be assessed using routine immunohistochemistry in participants from whom a muscle biopsy was obtained before and after surgery.
Change in biomarkers measured via blood samples after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  Blood samples will be taken to obtain plasma and serum in 6 mL tubes. Then, the samples will be centrifuged at 2500 rpm × 15 min. The plasma and serum will be distributed in microtubes and stored in a freezer at -80 °C until the evaluation by ELISA of the biomarkers (Cartilage remodeling: CTX-II and COMP; Bone remodeling: CTX-I and OC, and Muscle mass: PIIINP and SI) using Human Kits following the manufacturer's recommendations.
Change in functional capacity measured via Timed Up and Go test (TUG) after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before and after the 12-week intervention
  The functional capacity is assessed through the adapted Timed Up and Go test (TUG).
Change in muscle strength measured via 1RM strength tests after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention
  Maximum strength will be assessed according to 1RM strength tests on leg press, leg extension and leg abductor exercises (TuffStuff Fitness International, Los Angeles, USA), and on chest press, lat pulldown and horizontal row exercises (Ffit Tech, Viseu, Portugal). During a familiarization trial, proper lifting technique will be demonstrated and practiced. Maximum strength will be estimated using the multiplerepetition testing procedure. In an additional session, each participant's 1RM will be determined as described previously. Maximal handgrip strength will be measured three times with each hand using a Jamar® electronic handheld dynamometer (model Plus+, Patterson Medical, Cedarburg, WI, USA). The highest value using the stronger hand will be reported.
Change in body composition measured via dual-energy X-ray absorptiometry scanning after resistance exercise training | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention
  Body composition will be determined in all participants at baseline, before and after 2 weeks of prehabilitation/usual care and after 12 weeks of intervention. Whole-body and leg lean mass and fat mass will be determined by Dual Energy X-Ray Absorptiometry-DEXA (software GE Lunar enCORE) using the system's software GE Lunar enCORE. Weight will be recorded on a SECA® platform scale (Madison, WI, USA) with an accuracy of 0.1 kg and height will be measured to an accuracy of 0.5 cm using a stadiometer coupled to the scale. Waist circumference will be measured on exhalation at the midpoint between the lowest rib and the iliac crest on the right half of the body with a CESCORF retractable metric measuring tape with an accuracy of 1 cm (Porto Alegre, RS, Brazil).
Change in quality of life measured via SF-36 scale after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  Te SF-36 scale assesses overall health status and functioning by exploring eight health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.
Change in Independence in Activities of Daily Living via Lawton and Brody questionnaire after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  The Independence on Activities of Daily Living is assessed through the Lawton and Brody questionnaire.
Change in Cognitive Function measured via MoCA questionnaire after resistance exercise training. | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  The cognitive function is assessed through the MoCA questionnaire.
Change in Nutritional Status measured via Mini Nutritional Assessment and Malnutrition Universal Screening Tool after resistance exercise training. | The assessments will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  The Nutritional Status is assessed through the Mini Nutritional Assessment (MNA) and Malnutrition Universal Screening Tool.
Change in Perceived Hip Functionality measured via Harris Hip Score Questionnaire. | The assessment will be conducted 2 weeks and 48 hours before surgery and after 12-week intervention.
  The auto-perceived hip functionality is assessed through the Harris Hip Score questionnaire.
Change in habitual physical activity measured via Physical Activity Scale for Elderly (PASE) after resistance exercise training | The assessment will be conducted 2 weeks and 48 hours before surgery and after the 12-week intervention.
  The habitual physical activity is assessed through the PASE questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de La Frontera, Temuco, Cautin, Chile